CLINICAL TRIAL: NCT00455611
Title: Evaluation of the Effects of Intra-thoracic Positive Pressure Applicated With CPAP (Continuous Positive Airway Pressure) on Ventricular Function in Patients With Chronic Heart Failure: Modification Induced on Baroreflex Sensitivity
Brief Title: Effects of CPAP on Ventricular Function Modifications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled in the study
Sponsor: Ospedale S. Giovanni Bosco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: gbosco4
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2007-04

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; Continuous Positive Airway Pressure; Baroreflex; Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP (Continuous Positive Airway Pressure)

SUMMARY:
To assess modifications of ventricular function induced by CPAP (Continuous Positive Airway Pressure).

DETAILED DESCRIPTION:
There are still few studies on the effects of positive intra-thoracic pressure on ventricular function and spontaneous baroreflex sensitivity changes. Aim of the study is to evaluate, in patients with chronic heart failure with an ejection fraction < 40%, the modifications of ventricular function induced by CPAP (Continuos Positive Airway Pressure) application. All the measurament will be made in basal condition (without CPAP) and with CPAP administration at 10 cmH2O via an oro-nasal mask.

Echocardiograpich evaluation: morphologic and hemodynamic evaluation is obtained with an echocardiographic exmination. Left ventricular measurement will be assessed in M-mode, under two dimensional guide) according to American Society of Echocardiography guidelines. Left ventricular ejection fraction will be assessed with Simpson method.

Right ventricle morphology will be evaluated categorizing dimensions in a) normal, b) mild enlargement, c) severely increased and d) reduced. Right ventricle area will also be quantified in tele-diastole and in meso-sistole in apical 4 chamber and parasternal short-axis.

Baroreflex control of heart rate was assessed by "sequence method" analysis of continuous blood pressure recordings obtained in basal condition and during CPAP. Data obtained by non invasive assessment of arterial pressure will be analized and values of arterial systolic, diastolic pressure and pulsatory period for each cardiac cicle will be registered.

Assessment via "sequence method" is founded on identification, every 10 minutes, on sequences characterized by a progressive increase both in pressure both in RR interval or, conversely, by a progressive reduction of pressure and RR interval evaluated on 4 or more cardiac cicles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure
* Chronic heart failure
* Ejection fraction < 40%

Exclusion Criteria:

* Age < 18 years
* Permanent atrial fibrillation
* Infiltrative cardiomyopathy
* Mild/moderate chronic obstructive lung disease
* Chronic heart failure
* Diabetes mellitus
* Chronic kidney failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of modification of ventricular function and baroreflex sensitivity of heart rate after CPAP administration

CONTACTS AND LOCATIONS:
Overall Officials: Federico Olliveri, MD, Study Director — ospedale San Giovanni Bosco ASL4
Locations (1):
- Ospedale San Giovanni Bosco Medicina d'Urgenza, Turin, Piedmont, Italy